CLINICAL TRIAL: NCT06163703
Title: Strengthening Child Social-Emotional Functioning and Healthy Lifestyle Behaviors Through Parent-Based Prevention in Families Experiencing Major Stressors
Brief Title: Strengthening Child Social-Emotional and Lifestyle Health in Families Experiencing Stress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Nada Goodrum, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00123900; 5P20GM130420 (NIH)
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Child Behavior; Sedentary Behavior; Self-regulation; Parenting
MeSH Terms: conditions — Child Behavior; Sedentary Behavior; Self-Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will receive a 12-session parent-based prevention program based on Family Life Skills Triple P.
  Interventions: Behavioral: Family Life Skills Triple P
- Waitlist Control (No Intervention): Participants in the waitlist control arm will not receive any intervention during the clinical trial. They will be placed on a waitlist and then offered the intervention once post assessments are complete.

INTERVENTIONS:
Behavioral: Family Life Skills Triple P — The intervention is a 12-session program that combines parenting support with trauma-informed life skills coaching. It includes content related to positive parenting strategies, self-regulation, coping with emotions, effective communication, dealing with the past, and developing healthy habits.
  Arms: Intervention

SUMMARY:
This study evaluates feasibility and preliminary efficacy of a parent-based prevention program to promote social-emotional and lifestyle behavior health among 3- to 9-year-old children in families experiencing major stressors.

DETAILED DESCRIPTION:
Social-emotional difficulties and unhealthy lifestyle behaviors are prevalent among children in the U.S. and are associated with negative health outcomes. These challenges are even more pronounced among families who deal with major stressors, such as parental trauma history and mental health difficulties, parental chronic illness (e.g., HIV), parental substance use, economic disadvantage, and racial discrimination. The purpose of this study is to assess the feasibility, acceptability, and preliminary efficacy of a parent-based preventive intervention targeting parental self-regulation, stress reduction, and positive parenting, to promote child social-emotional and lifestyle behavior health, among families where the parents (a) have a child aged 3 to 9 years old, (b) have concerns about their child's behavior, mood, and/or lifestyle health, and (c) are experiencing major stressors. The intervention to be tested is based on Family Life Skills Triple P.

ELIGIBILITY:
Inclusion Criteria:

1. Child between the ages of 3-9 years
2. Parent/caregiver willing to engage in the intervention who

   * is at least 18 years of age
   * is primary caregiver or guardian for the participating child
   * has concerns about the child's mood, behavior, and/or lifestyle health
   * is experiencing two or more major stressors of the following: trauma history, mental health difficulties, living with HIV, racial discrimination, substance misuse, and/or financial strain
   * is English speaking.

Exclusion Criteria:

a. Parent or child has

* a significant cognitive disability, developmental delay, or pervasive developmental disorder
* active suicidal or homicidal ideation
* psychotic symptoms (active hallucinations, delusions, or impaired thought processes)
* ongoing family violence occurring within the home and/or active involvement of child protect services related to child maltreatment allegations.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Intervention acceptability | post-intervention (T2, Weeks 16-18)
  Assessed as parent-reported liking and approval of the intervention on a 5-point response scale and satisfaction with the intervention on a 4-point response scale, with higher scores indicating greater acceptability.
Intervention appropriateness | post-intervention (T2, Weeks 16-18)
  Assessed as parent-reported applicability and suitability of the intervention on a 5-point response scale, with higher scores indicating greater appropriateness.
Intervention feasibility--Implementability | post-intervention (T2, Weeks 16-18)
  Assessed as parent-reported ease of use and overall implementability of the intervention on a 5-point response scale, with higher scores indicating greater feasibility.
Intervention feasibility--Attendance | Weekly throughout intervention period (Weeks 1-17)
  Assessed as parent attendance at intervention sessions using weekly attendance logs
Trial-related feasibility--Recruitment capability | Continuously throughout recruitment period, up to 156 weeks
  Assessed as the proportion of eligible children who enroll in the study.
Trial-related feasibility--Retention | Continuously through study period (Weeks 1-30)
  Assessed as the proportion of enrolled children who remain in the study through the length of the intervention, with proportion who dropout and reasons for dropout also collected.
Child social-emotional difficulties: Problem behaviors | baseline (T1, Weeks 0-2); post-intervention (T2, Weeks 16-18); follow-up (T3, Week 30)
  Assessed as parent-reported frequency of child problematic behaviors on a 7-point response scale (higher scores indicate greater frequency).
Child social-emotional difficulties: Depression and anxiety symptoms | baseline (T1, Weeks 0-2); post-intervention (T2, Weeks 16-18); follow-up (T3, Week 30)
  Assessed as parent-reported frequency of child depression and anxiety symptoms on a 4-point response scale (higher scores indicate greater frequency).
Child social-emotional difficulties: Strengths and difficulties | baseline (T1, Weeks 0-2); post-intervention (T2, Weeks 16-18); follow-up (T3, Week 30)
  Assessed as parent-reported agreement with statements about child strengths and difficulties on a 3-point response scale (higher scores indicate greater endorsement).
Child physical activity | baseline (T1, Weeks 0-2); post-intervention (T2, Weeks 16-18); follow-up (T3, Week 30)
  Assessed as daily time spent sedentary and in various activity intensities using a wrist-worn accelerometer.
Child screen time | baseline (T1, Weeks 0-2); post-intervention (T2, Weeks 16-18); follow-up (T3, Week 30)
  Assessed as parent-reported average daily time spent engaging in screen time, including: watching TV; using a computer; gaming on a console or hand-held device; and using a tablet or smart phone for activities such as viewing videos, playing games, and browsing the internet.
Child sleep | baseline (T1, Weeks 0-2); post-intervention (T2, Weeks 16-18); follow-up (T3, Week 30)
  Assessed using a wrist-worn accelerometer to calculate nighttime sleep duration and using a validated measure of parent-reported child sleep-wake behaviors on a 6-point response scale, with lower scores indicating more problematic behaviors.

SECONDARY OUTCOMES:
Parenting practices | baseline (T1, Weeks 0-2); post-intervention (T2, Weeks 16-18); follow-up (T3, Week 30)
  Assessed as parent self-reported frequency of positive and negative parenting behaviors on a 5-point response scale, with higher subscale scores indicating greater frequency of the respective behaviors.
Parenting self-regulation | baseline (T1, Weeks 0-2); post-intervention (T2, Weeks 16-18); follow-up (T3, Week 30)
  Assessed as parent self-rated agreement with statements about self-regulation as a parent on a 7-point response scale, with higher scores indicating greater self-regulation.
Parenting stress | baseline (T1, Weeks 0-2); post-intervention (T2, Weeks 16-18); follow-up (T3, Week 30)
  Assessed as parent self-rated frequency and intensity of daily parenting hassles on a 4--point response scale, with higher scores indicating more frequent and intense hassles.

CONTACTS AND LOCATIONS:
Overall Officials: Nada M Goodrum, Ph.D., Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No